CLINICAL TRIAL: NCT01756417
Title: An Open-Label, Fixed Sequence, Single and Multiple Dose Study in Male and Female Subjects to Investigate the Potential for Pharmacokinetic and Pharmacodynamic Interaction Between Metformin and JNJ-28431754
Brief Title: A Study to Investigate Whether Pharmacokinetic and Pharmacodynamic Interactions Exist Between Metformin and Canagliflozin (JNJ-28431754) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013636; 28431754NAP1004 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin (JNJ-28431754); Metformin; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Metformin; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin + canagliflozin (JNJ-28431754) (Experimental): Each volunteer will receive a single dose of metformin on Day 1 followed by canagliflozin (JNJ-28431754) once daily on Days 4 to 7. On Day 8, volunteers will receive a single dose of canagliflozin in combination with a single dose of metformin.
  Interventions: Drug: Metformin; Drug: Canagliflozin (JNJ-28431754)

INTERVENTIONS:
Drug: Metformin — One 1,000 mg tablet of metformin taken orally (by mouth) on Day 1 and Day 8.
Drug: Canagliflozin (JNJ-28431754) — Four 25 mg tablets of canagliflozin (JNJ-28431754) taken orally on Days 4 through 8.
  Other Names: JNJ-28431754

SUMMARY:
The purpose of this study is to investigate whether there is a drug-drug interaction between multiple doses of canagliflozin (JNJ-28431754) and a single dose of metformin. The safety and tolerability of canagliflozin will also be assessed.

DETAILED DESCRIPTION:
This study is an open-label (all volunteers and study staff know the identity of the assigned treatment), fixed sequence (all volunteers receive the same medication on the same days), single and multiple-dose study to determine how metformin (a blood glucose-lowering agent used to treat patients with diabetes) affects the pharmacokinetics (ie, how the body affects the drug) and the pharmacodynamics (ie, how the drug affects the body) of canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus). The effect of canagliflozin on the pharmacokinetics and pharmacodynamics of metformin will also be evaluated. The study will consist of 3 phases: a screening phase, an open-label treatment phase, and an end-of-study (or follow-up) phase. Each volunteer will participate in the study for approximately 39 days.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have a Body Mass Index (BMI [weight (kg) / height (m)2]) between 18.5 and 35 kg/m2, inclusive
* Volunteers must be non-smokers or non-tobacco users

Exclusion Criteria:

- History of or currently active illness that the Investigator considers to be clinically significant and should exclude the volunteer from the study or that could interfere with the interpretation of the study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of canagliflozin (JNJ-28431754) | Up to Day 8
  Cmax (a measure of the body's exposure to canagliflozin [JNJ-28431754]) will be compared before and after administration of a single dose of metformin.
The area under the plasma concentration-time curve (AUC) for canagliflozin (JNJ-28431754) | Up to Day 8
  AUC (a measure of the body's exposure to canagliflozin [JNJ-28431754]) will be compared before and after administration of a single dose of metformin.
The maximum plasma concentration (Cmax) of metformin | Up to Day 8
  Cmax (a measure of the body's exposure to metformin will be compared before and after administration of multiple doses of canagliflozin (JNJ-28431754).
The area under the plasma concentration-time curve (AUC) for metformin | Up to Day 8
  AUC (a measure of the body's exposure to metformin will be compared before and after administration of multiple doses of canagliflozin (JNJ-28431754).
24-hour urine glucose excretion | Up to Day 10
  24-hour urine glucose excretion will be compared following a single dose of metformin, multiple doses of canagliflozin (JNJ-28431754), or multiple doses of canagliflozin in combination with a single dose of metformin.
24-hour area under the serum glucose concentration-time curve | Up to Day 8
  24-hour area under the serum glucose concentration-time curve will be compared following a single dose of metformin, multiple doses of canagliflozin (JNJ-28431754), or multiple doses of canagliflozin in combination with a single dose of metformin.

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Neptune City, New Jersey, United States

REFERENCES:
- See also: An Open-Label Study to Investigate the Absorption, Metabolism, and Excretion of JNJ-28431754 in Healthy Male Subjects Following a Single Oral Dose Administration of 14C-JNJ-28431754 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=2030&filename=CR013636_CSR.pdf